CLINICAL TRIAL: NCT00550667
Title: Clinical and Neuropsychological Validity of Attention-Deficit Hyperactivity Disorder in Adulthood
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200705065R
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention-deficit hyperactivity disorder; adult; diagnostic validity; neuropsychological functions; social functioning
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Social Adjustment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to establish the psychometric properties of the Adult ADHD Quality of Life Scale (AAQoL) and to validate the diagnosis of adult ADHD by ADHD symptoms, other clinical psychiatric symptoms, neuropsychological functioning, social/family/occupational functioning, and intervention effect.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a common (5-10%) childhood-onset neuropsychiatric disorder worldwide among children and adolescents with 50- 60% persistence to adulthood (3-4%). Western studies have revealed a wide range of family/social/occupational impairment and neurocognitive deficits in adults with ADHD. However, there is limited data on the treatment effect for adults with ADHD worldwide and there is lack of information about adult ADHD in Taiwan. In view of this, it is warranted to conduct a study on the clinical, functional, and neurocognitive aspects of adult ADHD in Taiwanese population.

This study consists of two parts: (1) a community survey among 1000 adults to establish the validity of AAQoL; and (2) a case-control study with a sample of 60 adults, aged 18-50, with DSM-IV ADHD and 60 healthy controls matching for the age and sex structure of the ADHD group. The instruments include a standard psychiatric diagnostic interviews using (K-SADS-E), self-administered rating scales for assessing psychopathology (ASRI), ADHD symptoms (ASRS, CGI-ADHD-S,), social and family functions (AAQoL, SDS, Moos dyadic assessment, family APGAR, GDS) and neuropsychological assessment (WAIS-III, CANTAB). The ADHD group will be reassessed for symptom severity and neuropsychological functioning 2-3 months (ranging from 8 to 12 weeks) after the first assessment.

We anticipate that this study will provide the primitive data on the symptomatology, neuropsychological functions, quality of life, and social/family function of adult patients with ADHD, will evaluate the treatment response of medication or psychosocial intervention in the aspects of symptomatology, neuropsychological functions, quality of life, and family function; and young psychiatric researchers will learn to conduct standardized psychiatric interview and neuropsychological tests, and to collect data, conduct statistical analysis, and prepare the manuscript. Our findings should have clinical implication in assessing and treating adult patients with ADHD and provide the preliminary data for future brain imaging, neurocognitive, and interventional studies on adult ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Case group:

Case group I: The cases with childhood ADHD diagnosis diagnosed as ADHD after interview Case group II: The cases with sufficient ADHD symptoms for diagnosis as DSM-IV ADHD at childhood but never assessed or treated for ADHD in childhood

* Control group：The subjects without the DSM-IV-TR diagnosis of ADHD or any major psychiatric disorders.

Exclusion Criteria:

* Comorbid with DSM-IV-TR diagnosis of pervasive developmental disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar affective disorder, severe anxiety disorder(such as OCD, ASD or PTSD) and mental retardation.
* In the major depressive episode, comorbid with severe anxiety disorders or during substance intoxication or withdrawal at the time of evaluation.
* With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy.
* With visual or hearing impairments, or motor disability which may influence the process of neuropsychological assessment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample & clinical sample
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Candido RCF, Menezes de Padua CA, Golder S, Junqueira DR. Immediate-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2021 Jan 18;1(1):CD013011. doi: 10.1002/14651858.CD013011.pub2. PMID 33460048
- [Derived] Ni HC, Shang CY, Gau SS, Lin YJ, Huang HC, Yang LK. A head-to-head randomized clinical trial of methylphenidate and atomoxetine treatment for executive function in adults with attention-deficit hyperactivity disorder. Int J Neuropsychopharmacol. 2013 Oct;16(9):1959-73. doi: 10.1017/S1461145713000357. Epub 2013 May 14. PMID 23672818